CLINICAL TRIAL: NCT00233818
Title: An Evaluation of Sirolimus-Coated Modified BX VELOCITY Balloon-Expandable Stents for the Treatment of Patients With de Novo Native Coronary Artery Lesions
Brief Title: FIM-NL - First-in-Man Study (Netherlands Part) With Sirolimus Coated Modified BX Velocity Stent
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC99-07
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Device: Sirolimus-coated Bx VELOCITY Stent

INTERVENTIONS:
Device: Sirolimus-coated Bx VELOCITY Stent

SUMMARY:
The objective of this study is to assess the performance and safety of a formulation of the antiproliferative agent, sirolimus coated on modified Bx VELOCITY Balloon-Expandable Stent mounted on the Raptor Over The Wire (OTW) Stent Delivery System (SDS) in patients with de novo coronary artery lesions.

DETAILED DESCRIPTION:
This is a single center, non-randomized study. Patients who meet the eligibility criteria will be treated with the sirolimus coated modified Bx VELOCITY Balloon-Expandable Stent mounted on the Raptor OTW SDS. Patients will be followed for five years post-procedure, with all patients having a repeat angiography at 6 months, 18 months, and 48 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS) or a positive ischemia study;
2. Single de novo lesion requiring treatment in a major native coronary artery;
3. Target lesion is <=18mm in length (visual estimate);
4. Target lesion is >=3.0mm and <=3.5mm in diameter (visual estimate);
5. Target lesion stenosis is >50% and <100% (visual estimate);

Exclusion Criteria:

1. A Q-wave or non-Q-wave myocardial infarction within the preceding 72 hours unless the CK and CK-MB enzymes are back to normal;
2. Unprotected left main coronary disease with >=50% stenosis;
3. Have an ostial target lesion;
4. Angiographic evidence of thrombus within target lesion;
5. Calcified lesions which cannot be successfully predilated;
6. Ejection fraction <=30%;
7. Target lesion involves bifurcation (either stenosis of both main vessel and major branch or stenosis of just major branch);
8. Totally occluded vessel;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-02; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Assessment of in-stent percent diameter stenosis (%DS) measured by quantitative coronary angiography. | post procedure and 6 months

SECONDARY OUTCOMES:
Assessment of lesion morphology by intravascular ultrasound (IVUS). | post procedure and 6 months
Target vessel failure (TVF). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, MD, Principal Investigator — Erasmus Centrum Thoraxcentrum
Locations (1):
- Erasmus Centrum Thoraxcentrum, Rotterdam, Netherlands

REFERENCES:
- [Result] Rensing BJ, Vos J, Smits PC, Foley DP, van den Brand MJ, van der Giessen WJ, de Feijter PJ, Serruys PW. Coronary restenosis elimination with a sirolimus eluting stent: first European human experience with 6-month angiographic and intravascular ultrasonic follow-up. Eur Heart J. 2001 Nov;22(22):2125-30. doi: 10.1053/euhj.2001.2892. PMID 11686669
- [Result] Degertekin M, Serruys PW, Foley DP, Tanabe K, Regar E, Vos J, Smits PC, van der Giessen WJ, van den Brand M, de Feyter P, Popma JJ. Persistent inhibition of neointimal hyperplasia after sirolimus-eluting stent implantation: long-term (up to 2 years) clinical, angiographic, and intravascular ultrasound follow-up. Circulation. 2002 Sep 24;106(13):1610-3. doi: 10.1161/01.cir.0000034447.02535.d5. PMID 12270850